CLINICAL TRIAL: NCT03197519
Title: Evaluation of a Treatment Program for Eating Disorders That Combines Face-to-face Cognitive Behavioural Treatment With an Online Intervention Using the TCapp Application, Within the Framework of Broader Research Project Entitled mHealth: Challenges and Opportunities for Health Systems
Brief Title: Evaluation of a Program for Eating Disorders That Combines Cognitive-behavioral Therapy With Online Psychological Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Oberta de Catalunya (Other)
Collaborators: La Caixa Foundation (Other)
Responsible Party: Principal Investigator, Francisco Lupiáñez Villanueva, Associate Professor and Researcher at the Faculty of Information and Communication Sciences, Universitat Oberta de Catalunya
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016ACUP 00056; TCApp.2017-01 (Other: Protocol ID assigned when protocol was submitted for approval to the Ethics Committees of the participating hospitals)
Record Dates: First submitted 2017-05-30; First posted 2017-06-23 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: mHealth; Eating Disorder
Keywords: mHealth; Eating Disorders; Randomised Controlled Trial; Cognitive Behavioural Therapy; cost effectiveness
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group will receive treatment as usual, that is to say, the standard treatment based on CBT principles that is offered by the different ED units in Spain, plus an online intervention using TCApp for a period of 12 weeks.
  Interventions: Behavioral: TCApp
- TAU control group (Other): The TAU control group will receive treatment as usual, offered by the different ED units in Spain. Patients from the control group will be offered access to TCApp after a 6-month period.
  Interventions: Behavioral: TAU

INTERVENTIONS:
Behavioral: TCApp — During these 12 weeks, in addition to TAU, the patient from the experimental group should use TCApp at least once a day, completing at least one self-record daily and/or contacting his/her therapist via chat when needed. The therapist responsible for the online monitoring should, at least once a week, connect to the online platform and perform the following actions: follow the patient's daily self-records, generate personalized reports or graphs and communicate with him/her via chat. After a 12-week period, patients from the experimental group and their therapists will stop using the TCApp application (they will be discharged).
  Arms: Experimental group
Behavioral: TAU — The TAU control group will receive treatment as usual, that is to say, the standard face-to-face CBT, offered by the different ED units in Spain.
  Arms: TAU control group

SUMMARY:
The purpose of this project is to conduct a multicentre, randomized controlled trial (RCT) with 250 patients diagnosed with an eating disorder (ED). In this experiment, the patients from the experimental group will test an mHealth application (TCApp developed by HealthApp) and then, a clinical efficacy analysis and economic evaluations will be performed. To do this, we have set the following three specific objectives:

* To evaluate the clinical efficacy of an intensive intervention that includes both standard face-to-face Cognitive Behavioural Treatment (CBT) (treatment as usual, TAU) plus an online intervention using TCApp, versus TAU alone.
* To carry out an economic evaluation (cost-utility and cost-effectiveness analysis) of the new mHealth intervention and identify factors that promote or hinder the implementation of TCApp in mental health settings in Spain.
* To analyse the adoption processes of this type of applications by patients and health professionals and identify the determinants of mHealth adoption.

General hypothesis:

The implementation of the intensive intervention program (TAU + TCApp) would result in a more significant improvement of the ED symptoms compared to the TAU control group.

Specific hypotheses:

* The application of the intensive mHealth intervention would lead to significantly greater change scores (difference between T0 and T1) in the primary outcome variable of ED psychopathology, compared to the control group.
* The mHealth intervention would lead to significantly greater change scores (difference between T0 and T1) in patients' secondary outcome variables: a) depression symptoms, b) anxiety symptoms, c) motivation to change, d) suicidal risk, and e) quality of life, compared to the control group.
* Similarly, intensive intervention would result in greater change scores (difference between T0 and T1) in caregivers' variables: a) quality of life and b) caregiver burden.

DETAILED DESCRIPTION:
1. The TCApp application TCapp is a tool intended to connect patients and therapists in the time between medical consultations. It is currently available on Google Play and Apple Store markets, there are more than 412 patients who are currently using it and it was developed in collaboration with different public and private mental health institutions in the Barcelona area (Althaia, Hospital de Sant Rafael, CST, ITA and Hospital Sant Joan de Déu). TCApp was designed from the start with therapists' and patients´ needs and interests in mind. By using TCapp, patients and therapists are in continuous contact, allowing for a quicker reaction from the therapist according to the patients' needs.

   With TCApp, patients can record their thoughts, behaviors, emotions and whatever the therapists consider relevant for the therapy, since the app can be customized according to the therapy requirements of each specific patient. It involves algorithms based on artificial intelligence that can generate alarms when strategic words (i.e. suicide, death, etc.) are written. It also introduces technologies that allow for real-time online contact with therapists and gamification aesthetics that include prizes, rewards and reminders aimed at improving patients' engagement.

   The BackOffice tool for therapists is a web-based platform where therapists can see in real time what their patients have registered (i.e. generation of graphs in a period of time to visualize parameter comparison and patient evolution) and they can interact in real time with them by using PUSH notifications. The tool is integrated in Azure server in order to ensure accordance with the most restrictive data protection laws and it is prepared for for its integration in the local management systems of hospitals and clinics. Finally, there is currently no application available to provide the same services and benefits as TCapp as most of the available applications contain self-help functionalities, rather than allowing for a bidirectional link between the patient and the therapist.

   Once TCApp has proven to be an efficient and effective tool for use in ED units of public and private mental health services in Spain, the long-term contributions of the current study are as follows:
   * To promote the clinical use of TCApp in ED units not only in Spain but also at an international level.
   * Reduce the direct and indirect costs associated with the treatment of eating disorders.
   * Improve the quality of patient care and the treatment effectiveness for EDs (e.g., increase patients' adherence to treatment, prevent relapse) while reducing waiting lists at various hospitals from Spain.
   * Explore the future export of the application to other mental disorders whose treatment is also based on cognitive behavioural therapy, such as depression, addictions and anxiety.
2. Work plan and duration of the project 2.1 Methods 2.1.1 Sample The total sample will include approximately 250 patients with an ED diagnosis currently receiving treatment, who will be recruited from different public and private mental health services in Spain (Parc Taulí Hospital, Sant Joan de Déu Hospital, Dexeus University Hospital of the Quirónsalud group in Barcelona, Sant Rafael Hospital, Servei Salut de les Illes Balears and Infantil Universitario Niño Jesús de Madrid). All patients will receive standard CBT treatment, which includes the support of a multidisciplinary team from the different ED units (psychiatry, psychology, nutrition, nursing).

The a priori sample size calculation was based on results from previous studies that implemented Internet-based programs in the treatment of EDs (Aardoom et al., 2013; Hötzel et al., 2014; Ruwaard et al., 2013). A small between-group effect size (Cohen' s d = 0.40) is expected. The calculation was conducted by the software program G*POWER. The primary analysis will concern the hypothesis that the average level of eating pathology at post-intervention in the control group, based on the EDE-Q scores, will be significantly higher than the average levels of eating pathology in the experimental group. Assuming an alpha of 0.05 and a power of 0.80 (β -1) in an independent samples one-way t-test, a minimum of 100 participants would be required per study arm. Allowing for a dropout rate of 25% of study participants from the baseline, 250 participants need to be recruited in total.

2.1.2 Design and procedure We will follow a mixed-methods approach, combining quantitative and qualitative methods, through a randomised controlled trial with an intensive intervention (TAU + TCApp) and a TAU control condition.

First, all material with information related to the study (research protocol, informed consent, patient information sheet, Data Collection Logbook, safety- and privacy-related issues concerning the TCApp application) will be submitted for approval to each one of the Ethical Committees of the participating hospitals. It should be mentioned that the approval of the Ethical Committee of the University leading the study (Universitat Oberta de Catalunya) was obtained on February 21st, 2017.

Participants will be recruited after previous recommendation by one of the ED specialists working at each centre. Specialists will do a preliminary screening taking into consideration the inclusion and exclusion criteria in order to identify potential candidates for the study. Interested individuals will be able to confirm their participation by notifying the ED specialist who will be responsible for their treatment. Then, an informational letter and an informed consent form will be delivered to them.

After completing and signing the informed consent form (for patients under 18 years of age, their parents will have to sign the informed consent), initial clinical interviews will be conducted by psychologists or other collaborators working in the ED unit. All the interviewers will be previously trained in administering the K-SADS-PL or SCID interview, depending on the participant's age. The objective of these interviews is: a) to definitively determine whether participants are eligible for the study according to the inclusion criteria, b) to establish the diagnosis for each patient and c) to evaluate them for possible comorbidities. At this time, sociodemographic and clinical data of each patient will also be collected through a brief interview. Then, those who meet the inclusion criteria will be invited to complete the baseline questionnaires for the study. During this baseline evaluation (T0), questionnaires will be administered to patients, their informal caregivers and the ED specialist responsible for the online monitoring of each patient. In addition, telephone interviews will be conducted with the technical staff and the ED specialists.

After completion of the baseline questionnaires, participants will be randomized to one of the two study conditions (experimental and control group). Randomization will be carried out by an independent researcher in blocks of 10 participants within each ED unit (50% of patients from each block will be assigned to the experimental group and the other 50% to the control group), using a random allocation program.

After this, patients will be notified about the group they belong to during their next visit to the ED unit. At this time, patients from the experimental group will be given oral and written instructions about how to download and use TCApp. In turn, patients from the TAU control group will be told that access to TCApp will be offered to them after a waiting period of 6 months.

Then, each group of patients will receive the treatment that corresponds to them during a period of 12 weeks. At the end of the 12-week treatment, patients from the experimental group will stop using TCApp and the evaluation post-treatment (T1, 12 weeks later) will be carried out and will include: a) a brief clinical interview (patients), b) questionnaires (patients, informal caregivers, ED specialists); c) telephone interviews (technical staff, ED specialists) and d) a focus groups with ED specialists of each institution who are interested in participating as well as with patients of the experimental group.

Both intent-to-treat and completers analyses will be carried out. Intent-to-treat analysis will include every participant who was randomly allocated to one of the study conditions, that is to say, 250 patients. Whenever possible, we will try to collect follow-up data from participants who have dropped out, in order to keep our dataset as complete as possible. Baseline differences between completers and dropouts will be analysed using data from the clinical interviews and the baseline questionnaires, and possible reasons for dropout will be examined through interviews with ED specialists (T1).

A participant will be considered a completer if he/she has completed the initial clinical interview as well as T0 and T1 evaluations. For participants from the experimental group to be considered completers, they will have to have used TCApp at least 70% of the time initially agreed upon before the start of the experiment (i.e., at least once a day during a period of 12 weeks). Only data from completers will be used to determine the treatment effect on the main outcome variable.

2.1.3 Study conditions The experimental group will receive the standard treatment based on CBT principles that is offered by the different ED units in Spain, plus an online intervention using TCApp for a period of 12 weeks. Only one ED specialist will be responsible for the online monitoring of each patient. For the specific purposes of our study, this role has been assigned to the nursing staff for most of the centres.

The TCApp application provides patients with a number of different functions, including daily self-records of their thoughts, emotions and behaviors, a chat with their therapists and motivational exercises. A TCApp online platform is also available for therapists for the online monitoring of each patient. Here, therapists have the possibility to follow the patient's daily self-records, generate personalized reports and graphs and communicate with him/her via chat, based on the information that the patient has provided online.

During these 12 weeks, the patient should use TCApp at least once a day, completing at least one self-record daily and/or contacting his/her therapist via chat when needed. The therapist responsible for the online monitoring should, at least once a week, connect to the online platform and perform the following actions: follow the patient's daily self-records, generate personalized reports or graphs and communicate with him/her via chat. After a 12-week period, patients from the experimental group and their therapists will stop using the TCApp application (they will be discharged).

The TAU control group will receive the standard face-to-face CBT, offered by the different ED units in Spain. Patients from the control group will be offered access to TCApp after a 6-month period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of an Eating or Feeding Disorder, based on: a) the Schedule for Affective Disorders and Schizophrenia-Present and Lifetime version (K-SADS-S-PL) (DSM-5 criteria) for minor patients or b) the Structural Clinical Interview for DSM-5 (SCID-5-RV) for adult patients. The diagnosis should be one of the following types: Anorexia Nervosa; Bulimia nervosa; Binge Eating Disorder; Other Specified Feeding or Eating Disorder: Atypical Anorexia Nervosa, Bulimia nervosa (of low frequency and/or limited duration), Binge-eating disorder (of low frequency and/or limited duration), purging disorder, night eating syndrome.
* Treatment regimen: Day Hospital or Ambulatory treatment, regardless of the illness duration or the severity of the disorder
* Treatment received by ED unit of reference: Standard Cognitive Behavioural Therapy
* Understanding of Spanish, Catalan or English language, depending on the language option chosen by the participant for the TCApp
* Minimal digital skills and availability of proper mobile phone for patients

Exclusion Criteria:

* Age less than 12 years
* Treatment regimen: Hospitalization
* Diagnosis of psychosis
* Intellectual disability
* Have a mobile phone with a Windows Phone operating system

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2017-09-04 (Actual); Primary Completion 2018-09-07 (Actual); Study Completion 2018-09-07 (Actual)

PRIMARY OUTCOMES:
Change in Eating Disorder symptomatology I (patients) | Baseline-3 months
  Change from baseline assessment to 3 months assessment
Change in Eating Disorder symptomatology II (patients) | Baseline-3 months
  Change from baseline assessment to 3 months assessment in patient total score on Short Evaluation of Eating Disorders (SEED) (Bauer, Winn, Schmidt, & Kordy, 2005)

SECONDARY OUTCOMES:
Change in Depression (patients) | Baseline-3 months
  Change from baseline assessment to 3 months assessment
Change in Anxiety (patients) | Baseline-3 months
  Change from baseline assessment to 3 months assessment in patient total score on State-Trait Anxiety Inventory (STAI) (Spielberger, Gorsuch, Lushene, Vagg, & Jacobs, 1983)
Change in Motivation to change (AN patients) | Baseline-3 months
  Change from baseline assessment to 3 months assessment
Change in Treatment drop-out (patients) | Baseline-3 months
  Change from baseline to 3 months in number of patients who dropout based on healthcare professional statements (Yes or No), using a phone interview
Change in Suicide risk (patients) | Baseline-3 months
  Change from baseline assessment to 3 months assessment
Change in Quality of life (patients) | Baseline-3 months
  Change from baseline assessment to 3 months assessment in patient total score on EuroQoL-EQ-5D (Group EQ, 1990)
Change in Motivation to change (BN/BED/OSFED patients) | Baseline-3 months
  Change from baseline assessment to 3 months assessment in patient total score on Bulimia Nervosa Stages of Change Questionnaire (BNSOCQ) (Martínez, Castro, Bigorra, Morer, Calvo, Vila, Toro, & Riegel, 2007)

OTHER OUTCOMES:
Change in Caregiver burden (caregivers) | Baseline-3 months
  Change from baseline assessment to 3 months assessment
Change in Caregiver quality of life (caregivers) | Baseline-3 months
  Change from baseline assessment to 3 months assessment in caregiver total score on EuroQoL-EQ-5D (Group EQ, 1990)
Cost of mobile app development (TCApp) | Baseline
  Technical staff responses, using a phone interview (cost-effectiveness analysis)
Change in consumption of health resources, drugs consumption and school or work absenteeism (patients) | Baseline-3 months
  Change from baseline assessment to 3 months assessment in patient total score on iMTA Questionnaire: Healthcare consumption, illness and work associated with psychiatric illness (TiC-P) (cost-effectiveness analysis)
Change in consumption of health resources (patient) | Baseline-3 months
  Change from baseline assessment to 3 months assessment on the total number of visits with the ED specialist and with the emergency services based on the healthcare professional responses, using a phone interview (cost-effectiveness analysis)
Change in the amount of work (healthcare professionals) | Baseline-3 months
  Change from baseline assessment to 3 months assessment in the amount of working hours per day, also considering the pay rate per hour and the time dedicated to the online follow-up of each patient. This information will be collected through a phone interview (cost-effectiveness analysis)
Usability (TCApp) | 3 months
  ED specialist total score on System Usability Scale (SUS) (Broooke, 1986)
Usability (TCApp) | 3 months
  Patient total score on System Usability Scale (SUS) (Broooke, 1986)
Satisfaction (TCApp) | 3 months
  ED specialist total score on Client Satisfaction Questionnaire (CSQ-8) (Larsen et al., 1979)
Satisfaction (TCApp) | 3 months
  Patient total score on Client Satisfaction Questionnaire (CSQ-8) (Larsen et al., 1979)
Cost of mobile app maintenance (TCApp) | 3 months
  Technical staff responses, using a phone interview (cost-effectiveness analysis)
Change in consumption of health resources, drugs consumption and work absenteeism (caregivers) | Baseline-3 months
  Change from baseline assessment to 3 months assessment
Change in consumption of drugs (patient) | Baseline-3 months
  Change from baseline assessment to 3 months assessment in the consumption of drugs, based on the healthcare professional responses, using a phone interview (cost-effectiveness analysis)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Lupiañez Villanueva, PhD, Principal Investigator — Universitat Oberta de Catalunya
Locations (4):
- Spain (4):
  - Hospital Sant Joan de Déu, Barcelona
  - Hospital Universitario Dexeus del grupo Quirónsalud de Barcelona, Barcelona
  - Servei de Salut de les Illes Balears, Palma de Mallorca
  - Hospital Parc Taulí, Sabadell

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stuhldreher N, Konnopka A, Wild B, Herzog W, Zipfel S, Lowe B, Konig HH. Cost-of-illness studies and cost-effectiveness analyses in eating disorders: a systematic review. Int J Eat Disord. 2012 May;45(4):476-91. doi: 10.1002/eat.20977. Epub 2012 Feb 1. PMID 22294558
- [Background] Steinhausen HC. The outcome of anorexia nervosa in the 20th century. Am J Psychiatry. 2002 Aug;159(8):1284-93. doi: 10.1176/appi.ajp.159.8.1284. PMID 12153817
- [Background] Anastasiadou D, Medina-Pradas C, Sepulveda AR, Treasure J. A systematic review of family caregiving in eating disorders. Eat Behav. 2014 Aug;15(3):464-77. doi: 10.1016/j.eatbeh.2014.06.001. Epub 2014 Jun 19. PMID 25064301
- [Background] Fairburn CG, Rothwell ER. Apps and eating disorders: A systematic clinical appraisal. Int J Eat Disord. 2015 Nov;48(7):1038-46. doi: 10.1002/eat.22398. Epub 2015 Feb 27. PMID 25728705
- [Background] Bauer S, Moessner M. Harnessing the power of technology for the treatment and prevention of eating disorders. Int J Eat Disord. 2013 Jul;46(5):508-15. doi: 10.1002/eat.22109. PMID 23658102
- [Background] Loucas CE, Fairburn CG, Whittington C, Pennant ME, Stockton S, Kendall T. E-therapy in the treatment and prevention of eating disorders: A systematic review and meta-analysis. Behav Res Ther. 2014 Dec;63:122-31. doi: 10.1016/j.brat.2014.09.011. Epub 2014 Oct 5. PMID 25461787
- [Background] Jacobi C, Volker U, Trockel MT, Taylor CB. Effects of an Internet-based intervention for subthreshold eating disorders: a randomized controlled trial. Behav Res Ther. 2012 Feb;50(2):93-9. doi: 10.1016/j.brat.2011.09.013. Epub 2011 Nov 15. PMID 22137366
- [Background] Kass AE, Trockel M, Safer DL, Sinton MM, Cunning D, Rizk MT, Genkin BH, Weisman HL, Bailey JO, Jacobi C, Wilfley DE, Taylor CB. Internet-based preventive intervention for reducing eating disorder risk: A randomized controlled trial comparing guided with unguided self-help. Behav Res Ther. 2014 Dec;63:90-8. doi: 10.1016/j.brat.2014.09.010. Epub 2014 Oct 2. PMID 25461783
- [Background] Stice E, Durant S, Rohde P, Shaw H. Effects of a prototype Internet dissonance-based eating disorder prevention program at 1- and 2-year follow-up. Health Psychol. 2014 Dec;33(12):1558-67. doi: 10.1037/hea0000090. Epub 2014 Jul 14. PMID 25020152
- [Background] Aardoom JJ, Dingemans AE, Spinhoven P, Van Furth EF. Treating eating disorders over the internet: a systematic review and future research directions. Int J Eat Disord. 2013 Sep;46(6):539-52. doi: 10.1002/eat.22135. Epub 2013 May 15. PMID 23674367
- [Background] Schlegl S, Burger C, Schmidt L, Herbst N, Voderholzer U. The potential of technology-based psychological interventions for anorexia and bulimia nervosa: a systematic review and recommendations for future research. J Med Internet Res. 2015 Mar 31;17(3):e85. doi: 10.2196/jmir.3554. PMID 25840591
- [Background] Juarascio AS, Manasse SM, Goldstein SP, Forman EM, Butryn ML. Review of smartphone applications for the treatment of eating disorders. Eur Eat Disord Rev. 2015 Jan;23(1):1-11. doi: 10.1002/erv.2327. Epub 2014 Oct 10. PMID 25303148
- [Background] Nitsch M, Dimopoulos CN, Flaschberger E, Saffran K, Kruger JF, Garlock L, Wilfley DE, Taylor CB, Jones M. A Guided Online and Mobile Self-Help Program for Individuals With Eating Disorders: An Iterative Engagement and Usability Study. J Med Internet Res. 2016 Jan 11;18(1):e7. doi: 10.2196/jmir.4972. PMID 26753539
- [Background] Tregarthen JP, Lock J, Darcy AM. Development of a smartphone application for eating disorder self-monitoring. Int J Eat Disord. 2015 Nov;48(7):972-82. doi: 10.1002/eat.22386. Epub 2015 Jul 27. PMID 26213130
- [Background] Juarascio AS, Goldstein SP, Manasse SM, Forman EM, Butryn ML. Perceptions of the feasibility and acceptability of a smartphone application for the treatment of binge eating disorders: Qualitative feedback from a user population and clinicians. Int J Med Inform. 2015 Oct;84(10):808-16. doi: 10.1016/j.ijmedinf.2015.06.004. Epub 2015 Jun 15. PMID 26113461
- [Derived] Anastasiadou D, Lupianez-Villanueva F, Fauli C, Arcal Cunillera J, Serrano-Troncoso E. Cost-effectiveness of the mobile application TCApp combined with face-to-face CBT treatment compared to face-to-face CBT treatment alone for patients with an eating disorder: study protocol of a multi-centre randomised controlled trial. BMC Psychiatry. 2018 May 2;18(1):118. doi: 10.1186/s12888-018-1664-4. PMID 29716580